CLINICAL TRIAL: NCT03247530
Title: Evaluation of SPN-812 (Viloxazine Extended-release Capsule) 100 and 200 mg Efficacy and Safety in Children With ADHD - A Double-Blind, Placebo-Controlled, Pivotal Trial
Brief Title: Evaluation of SPN-812 (Viloxazine Extended-release Capsule) Low Dose in Children With ADHD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Supernus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 812P301
Record Dates: First submitted 2017-08-09; First posted 2017-08-11 (Actual); Results first posted 2021-06-02 (Actual); Last update posted 2021-07-02 (Actual); Status verified 2021-06

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Placebo, qd, oral capsule
  Interventions: Drug: Placebo
- 100mg SPN-812 (Experimental): 100mg SPN-812, qd, oral capsule
  Interventions: Drug: 100mg SPN-812
- 200mg SPN-812 (Experimental): 200mg SPN-812, qd, oral capsule
  Interventions: Drug: 200mg SPN-812

INTERVENTIONS:
Drug: Placebo — Placebo was administered once daily
  Other Names: PBO
  Arms: Placebo
Drug: 100mg SPN-812 — 100mg SPN-812 was administered once daily and compared to placebo
  Other Names: SPN-812
  Arms: 100mg SPN-812
Drug: 200mg SPN-812 — 200mg SPN-812 was administered once daily and compared to placebo
  Other Names: SPN-812
  Arms: 200mg SPN-812

SUMMARY:
This study will evaluate the efficacy and safety of low doses of SPN-812 in children 6-11 years of age diagnosed with ADHD.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled, 3-arm, parallel-group study, to assess the efficacy and safety of SPN-812 as monotherapy for the treatment of children 6-11 years old with ADHD.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy male or female subjects, 6-11 years of age, inclusive.
2. Diagnosis of ADHD according to the Diagnostic and Statistical Manual of Mental Disorders-5 (DSM-5), confirmed with the Mini International Neuropsychiatric Interview for Children and Adolescents (MINI-KID).
3. Attention Deficit/Hyperactivity Disorder Rating Scale-5, Home Version: Child, Investigator Administered and Scored (ADHD-RS-5) score of at least 28.
4. CGI-S score of at least 4 at screening.
5. Weight of at least 20 kg.
6. Free of medication for the treatment of ADHD for at least one week prior to randomization and agreement to remain so throughout the study.
7. Considered medically healthy by the Investigator via assessment of physical examination, medical history, clinical laboratory tests, vital signs, and electrocardiogram.
8. Written informed consent obtained from the subject's parent or legal representative and informed assent from the subject, if applicable.
9. Females of childbearing potential (FOCP) must be either sexually inactive (abstinent) or, if sexually active, must agree to use one of the following acceptable birth control methods beginning 30 days prior to the first dose, throughout the study:

   1. simultaneous use of male condom and intra-uterine contraceptive device placed at least four weeks prior to the first study drug administration
   2. surgically sterile male partner
   3. simultaneous use of male condom and diaphragm with spermicide
   4. established hormonal contraceptive

Exclusion Criteria:

1. Current diagnosis of major psychiatric disorders. Subjects with Major Depressive Disorder are allowed in the study if the subject is free of episodes both currently and for the last six months.
2. Current diagnosis of major neurological disorders. Subjects with seizures or a history of seizure disorder within the immediate family (siblings, parents), or a history of seizure-like events are excluded from the study.
3. Current diagnosis of significant systemic disease.
4. Evidence of suicidality (defined as either active suicidal plan/intent or active suicidal thoughts, or more than one lifetime suicide attempt) within the six months before Screening or at Screening.
5. BMI greater than 95th percentile for the appropriate age and gender.
6. History of an allergic reaction to viloxazine or related drugs.
7. Any food allergy, intolerance, restriction or special diet that, in the opinion of the Investigator, could contraindicate the subject's participation in this study.
8. Subjects who received any investigational drug within the longer of 30 days or 5 half-lives prior to Day 1 dosing of SM.
9. Any reason, which, in the opinion of the Investigator, would prevent the subject from participating in the study.
10. Positive drug screen at the Screening Visit. A positive test for amphetamines is allowed for subjects receiving a stimulant ADHD medication at Screening; the subject will be required to discontinue the stimulant for the study, beginning at least one week prior to the Baseline Visit.
11. Pregnancy or refusal to practice abstinence or acceptable birth control during the study (for female subjects of childbearing potential).

Ages: 6 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 477 (Actual)
Dates: Start 2017-10-20 (Actual); Primary Completion 2018-09-12 (Actual); Study Completion 2018-09-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stefan Schwabe, MD, Study Director — Supernus Pharmaceuticals, Inc.
Locations (7):
- United States (7):
  - Harmonex Neuroscience Research, Dothan, Alabama
  - Indago Research & Health Center, Inc., Hialeah, Florida
  - Advanced Clinical Research, Meridian, Idaho
  - Finger Lakes Clinical Research, Rochester, New York
  - Houston Clinical Trials, Houston, Texas
  - Family Psychiatry of the Woodlands, The Woodlands, Texas
  - Aspen Clinical Research, Orem, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Faraone SV, Gomeni R, Hull JT, Busse GD, Lujan B, Rubin J, Nasser A. Response of peer relations and social activities to treatment with viloxazine extended-release capsules (Qelbree(R) ): A post hoc analysis of four randomized clinical trials of children and adolescents with attention-deficit/hyperactivity disorder. Brain Behav. 2023 Apr;13(4):e2910. doi: 10.1002/brb3.2910. Epub 2023 Feb 27. PMID 36847750
- [Derived] Faraone SV, Gomeni R, Hull JT, Busse GD, Melyan Z, Rubin J, Nasser A. Executive Function Outcome of Treatment with Viloxazine Extended-Release Capsules in Children and Adolescents with Attention-Deficit/Hyperactivity Disorder: A Post-Hoc Analysis of Four Randomized Clinical Trials. Paediatr Drugs. 2021 Nov;23(6):583-589. doi: 10.1007/s40272-021-00470-2. Epub 2021 Sep 15. PMID 34523063
- [Derived] Nasser A, Kosheleff AR, Hull JT, Liranso T, Qin P, Busse GD, Fava M, Maletic V, Rubin J, Lopez F. Evaluating the likelihood to be helped or harmed after treatment with viloxazine extended-release in children and adolescents with attention-deficit/hyperactivity disorder. Int J Clin Pract. 2021 Aug;75(8):e14330. doi: 10.1111/ijcp.14330. Epub 2021 May 26. PMID 33971070
- [Derived] Nasser A, Kosheleff AR, Hull JT, Liranso T, Qin P, Busse GD, O'Neal W, Fava M, Faraone SV, Rubin J. Translating Attention-Deficit/Hyperactivity Disorder Rating Scale-5 and Weiss Functional Impairment Rating Scale-Parent Effectiveness Scores into Clinical Global Impressions Clinical Significance Levels in Four Randomized Clinical Trials of SPN-812 (Viloxazine Extended-Release) in Children and Adolescents with Attention-Deficit/Hyperactivity Disorder. J Child Adolesc Psychopharmacol. 2021 Apr;31(3):214-226. doi: 10.1089/cap.2020.0148. Epub 2021 Feb 17. PMID 33600233
- [Derived] Nasser A, Liranso T, Adewole T, Fry N, Hull JT, Chowdhry F, Busse GD, Cutler AJ, Jones NJ, Findling RL, Schwabe S. A Phase III, Randomized, Placebo-controlled Trial to Assess the Efficacy and Safety of Once-daily SPN-812 (Viloxazine Extended-release) in the Treatment of Attention-deficit/Hyperactivity Disorder in School-age Children. Clin Ther. 2020 Aug;42(8):1452-1466. doi: 10.1016/j.clinthera.2020.05.021. Epub 2020 Jul 25. PMID 32723670

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Placebo oral capsule
  Treatment A: Placebo oral capsule was administered once daily
- 100mg SPN-812: SPN-812 oral capsule
  Treatment B: 100mg SPN-812 was administered once daily and compared to placebo
- 200mg SPN-812: SPN-812 oral capsule
  Treatment C: 200mg SPN-812 was administered once daily and compared to placebo
Period: Overall Study
Arm/Group | Placebo | 100mg SPN-812 | 200mg SPN-812
Started (Number of subjects is based on the Safety Population (defined as subjects who were randomized and took at least one dose of study medication)) | 159 | 154 | 161
Completed | 132 | 126 | 141
Not Completed | 27 | 28 | 20
Not completed — Withdrawal by caregiver | 19 | 8 | 10
Not completed — Lost to Follow-up | 3 | 9 | 6
Not completed — Adverse Event | 2 | 5 | 2
Not completed — Failure to follow procedure | 1 | 1 | 1
Not completed — Withdrawal by Subject | 1 | 1 | 0
Not completed — Study medication misuse | 0 | 1 | 0
Not completed — Other, multiple categories | 1 | 3 | 1

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population: The ITT population includes subjects who were randomized, took at least one dose of study medication, have a baseline Attention-Deficit/Hyperactivity Disorder Rating Scale, 5th Edition (ADHD-RS-5) assessment and have at least one post-baseline ADHD-RS-5 assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | 100mg SPN-812 | 200mg SPN-812 | Total
Number analyzed (Participants) | 155 | 147 | 158 | 460
Age, Continuous [Mean (Standard Deviation); unit: years] | 8.5 (1.74) | 8.5 (1.70) | 8.5 (1.67) | 8.5 (1.70)
Age, Customized [Count of Participants; unit: Participants]
  6 to 9 years | 103 | 103 | 107 | 313
  10 to 11 years | 52 | 44 | 51 | 147
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 58 | 53 | 59 | 170
  Male | 97 | 94 | 99 | 290
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 32 | 38 | 51 | 121
  Not Hispanic or Latino | 123 | 108 | 107 | 338
  Unknown or Not Reported | 0 | 1 | 0 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 1 | 0 | 2
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 69 | 63 | 69 | 201
  White | 77 | 76 | 83 | 236
  More than one race | 7 | 7 | 6 | 20
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 155 | 147 | 158 | 460
ADHD-RS-5 Total Score [Mean (Standard Deviation); unit: units on a scale] — The Attention-Deficit/Hyperactivity Disorder Rating Scale, 5th Edition (ADHD-RS-5) is an ADHD-specific rating scale designed and validated to assess current ADHD symptomatology. It consists of 18 items that correspond to the 18 ADHD symptoms per the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5). Each item is rated on a 4-point Likert-type scale from 0 (never or rarely) to 3 (very often). Total score = sum of 18 items (range: 0 to 54). The higher the score, the more severe the ADHD symptoms (a total score >=28 was an inclusion criterion of this study).
  units on a scale | 43.6 (7.05) | 45.0 (6.53) | 44.0 (6.80) | 44.2 (6.81)
ADHD-RS-5 Inattention Subscale Score [Mean (Standard Deviation); unit: units on a scale] — The Attention-Deficit/Hyperactivity Disorder Rating Scale, 5th Edition (ADHD-RS-5) is an ADHD-specific rating scale designed and validated to assess current ADHD symptomatology. It consists of 18 items that correspond to 18 ADHD symptoms per DSM-5, including 9 items for the Hyperactivity/Impulsivity (HI) subscale and 9 items for the Inattention (IA) subscale. Each item is rated on a 4-point Likert-type scale from (0=never or rarely to 3=very often). The IA Subscale score = sum of all 9 IA items on the ADHD-RS-5 (range: 0 to 27). The higher the score, the more severe the IA symptoms of ADHD.
  units on a scale | 22.5 (3.79) | 22.8 (3.24) | 22.9 (3.53) | 22.7 (3.53)
ADHD-RS-5 Hyperactivity/Impulsivity Subscale Score [Mean (Standard Deviation); unit: units on a scale] — The Attention-Deficit/Hyperactivity Disorder Rating Scale, 5th Edition (ADHD-RS-5) is an ADHD-specific rating scale designed and validated to assess current ADHD symptomatology. It consists of 18 items that correspond to 18 ADHD symptoms per DSM-5, including 9 items for the Hyperactivity/Impulsivity (HI) subscale and 9 items for the Inattention (IA) subscale. Each item is rated on a 4-point Likert-type scale (0=never or rarely to 3=very often). The HI Subscale score = the sum of all 9 HI items on the ADHD-RS-5 (range: 0 to 27). The higher the score, the more severe the HI symptoms of ADHD.
  units on a scale | 21.1 (4.90) | 22.2 (4.65) | 21.1 (5.15) | 21.5 (4.92)

OUTCOME MEASURES:

1. Primary Outcome: Efficacy of SPN-812 Assessed by Attention-Deficit/Hyperactivity Disorder (ADHD) Rating Scale, 5th Edition (ADHD-RS-5)
Description: The Primary Endpoint was the change from baseline in the Attention-Deficit/Hyperactivity Disorder Rating Scale, 5th Edition (ADHD-RS-5) Total score at Week 6 (End of Study). The ADHD-RS-5 is an ADHD-specific rating scale designed and validated to assess current ADHD symptomatology. The scale consists of 18 items that directly correspond to the 18 Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5) symptoms of ADHD. Each item is rated on a 4-point Likert-type scale from 0 (never or rarely) to 3 (very often). A Total score is calculated by adding the responses of all 18 items (range: 0-54; the higher the score, the more severe the ADHD symptoms). Lower change from baseline scores (<0) represent a better outcome.
Time Frame: Baseline and Week 6 (End of Study)
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- Placebo: Placebo, oral capsule
  Treatment A: Placebo was administered once daily
Arm/Group | Placebo | 100mg SPN-812 | 200mg SPN-812
Number analyzed (Participants) | 155 | 147 | 158
score on a scale | -10.9 (1.14) | -16.6 (1.16) | -17.7 (1.12)
Statistical Analysis 1: Comparison: Placebo vs 100mg SPN-812; Test type: Superiority; p = 0.0004, Mixed Models for Repeated Measures; Least Square Mean Difference = -5.8, 95% CI 2-sided [-8.9 to -2.6], Standard Error of Mean 1.61
Statistical Analysis 2: Comparison: Placebo vs 200mg SPN-812; Test type: Superiority; p < 0.0001, Mixed Models for Repeated Measures; Least Square Mean Difference = -6.9, 95% CI 2-sided [-10.0 to -3.8], Standard Error of Mean 1.58

2. Secondary Outcome: Effect of SPN-812 Assessed by Clinical Global Impression-Improvement (CGI-I) Scale
Description: The first Key Secondary Endpoint was the Clinical Global Impression-Improvement (CGI-I) Scale score at Week 6 (End of Study). The CGI-I scale is a single item assessment of how much the patient's illness has improved or worsened relative to a baseline state prior to the beginning of treatment. The CGI-I is rated on a 7-point Likert scale from 1 to 7, where 1 = "very much improved" and 7 = "very much worse." Successful therapy is indicated by a lower overall score in subsequent testing.
Time Frame: Week 6 (End of Study)
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Groups:
- 200mg SPN-812: SPN-812, oral capsule
  Treatment C: 200mg SPN-812 was administered once daily and compared to placebo
Arm/Group | Placebo | 100mg SPN-812 | 200mg SPN-812
Number analyzed (Participants) | 155 | 147 | 158
score on a scale | 3.1 (0.10) | 2.7 (0.10) | 2.6 (0.09)
Statistical Analysis 1: Comparison: Placebo vs 100mg SPN-812; Test type: Superiority; p = 0.0020, ANCOVA; ANCOVA model with baseline Clinical Global Impression-Severity of Illness (CGI-S) score and treatment as fixed independent variables; Mean Difference (Final Values) = -0.4, 95% CI 2-sided [-0.7 to -0.2], Standard Error of Mean 0.14
Statistical Analysis 2: Comparison: Placebo vs 200mg SPN-812; Test type: Superiority; p < 0.0001, ANCOVA; [statistical method as in outcome 2, analysis 1]; Mean Difference (Final Values) = -0.6, 95% CI 2-sided [-0.8 to -0.3], Standard Error of Mean 0.13

3. Secondary Outcome: Effect of SPN-812 Assessed by Conners 3 - Parent Short Form (C3PS)
Description: The second Key Secondary Endpoint was the change from baseline in the Conners 3rd Edition - Parent Short Form (C3PS) Composite T-score at Week 6 (End of Study). The Conners 3rd Edition is a focused diagnostic tool for the assessment of ADHD and associated learning, behavior, and emotional problems in children 6 to 18 years of age. The C3PS is completed by a child's parent/guardian and is comprised of 45 items with subsets of items related to six content scales: inattention, hyperactivity/impulsivity, executive functioning, learning problems, defiance/aggression and peer relations. The parent rates his/her child on the first 43 items of the C3PS using a 4-point Likert scale (0-3; where 0=not at all true [never, seldom] and 3=very much true [very often, very frequently]) based on past month; the last 2 items are fill-in-the-blank and do not contribute to the raw score(s). Raw scores are converted to T-scores. Lower change from baseline T-scores (<0) represent a better outcome.
Time Frame: Baseline and Week 6 (End of Study)
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Placebo | 100mg SPN-812 | 200mg SPN-812
Number analyzed (Participants) | 155 | 147 | 158
T-score | -4.8 (0.81) | -9.1 (0.83) | -9.2 (0.82)
Statistical Analysis 1: Comparison: Placebo vs 100mg SPN-812; Test type: Superiority; p = 0.0003, ANCOVA; Mean Difference (Final Values) = -4.2, 95% CI 2-sided [-6.5 to -1.9], Standard Error of Mean 1.16
Statistical Analysis 2: Comparison: Placebo vs 200mg SPN-812; Test type: Superiority; p = 0.0002, ANCOVA; Mean Difference (Final Values) = -4.3, 95% CI 2-sided [-6.6 to -2.1], Standard Error of Mean 1.15

4. Secondary Outcome: Effect of SPN-812 Assessed by Weiss Functional Impairment Rating Scale-Parent Report (WFIRS-P)
Description: The third Key Secondary Endpoint was the change from baseline in the Weiss Functional Impairment Rating Scale-Parent Report (WFIRS-P) Total Average score at Week 6 (End of Study). The WFIRS instrument evaluates ADHD-related functional impairment. The WFIRS-P is completed by the child's parent/guardian and is comprised of 50 items grouped into six domains: Family (10 items), School (10 items, includes learning [4 items] and behavior [6 items]), Life Skills (10 items), Child's Self-Concept (3 items), Social Activities (7 items), and Risky Activities (10 items). The parent/guardian rates each item on a 4-point Likert scale (0-3; where 0=never or not at all to 3= very often or very much) based on their child's behavior past month. A Total Average score was computed by calculating mean rating of all 50 items (ranging from 0 to 3, where a higher value represents more severe functional impairment). Lower change from baseline Total Average scores (<0) represent a better outcome.
Time Frame: Baseline and Week 6 (End of Study)
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | 100mg SPN-812 | 200mg SPN-812
Number analyzed (Participants) | 155 | 147 | 158
score on a scale | -0.22 (0.033) | -0.36 (0.033) | -0.39 (0.032)
Statistical Analysis 1: Comparison: Placebo vs 100mg SPN-812; Test type: Superiority; p = 0.0019, ANCOVA; Least Square Mean Difference = -0.14, 95% CI 2-sided [-0.24 to -0.05], Standard Error of Mean 0.047
Statistical Analysis 2: Comparison: Placebo vs 200mg SPN-812; Test type: Superiority; p = 0.0020, ANCOVA; Least Square Mean Difference = -0.17, 95% CI 2-sided [-0.26 to -0.08], Standard Error of Mean 0.046

5. Secondary Outcome: Effect of SPN-812 Assessed by 50% Responder Rate Per the Attention-Deficit/Hyperactivity Disorder Rating Scale, 5th Edition (ADHD-RS-5)
Description: An additional secondary endpoint was the percentage of responders at Week 6 (End of Study). A responder was defined as a subject who had a 50% or greater reduction (improvement) in their change from baseline Attention-Deficit/Hyperactivity Disorder Rating Scale, 5th Edition (ADHD-RS-5) Total score at Week 6 (End of Study). Values range from 0 to 100%. A higher percentage represents a greater number of responders.
Time Frame: Week 6 (End of Study)
Population: as for baseline characteristics
Measure: Number; unit: percentage of subjects
Groups:
- Placebo: Placebo oral capsule
  Treatment A: Placebo was administered once daily
Arm/Group | Placebo | 100mg SPN-812 | 200mg SPN-812
Number analyzed (Participants) | 155 | 147 | 158
percentage of subjects | 19.8 | 34.2 | 41.2
Statistical Analysis 1: Comparison: Placebo vs 100mg SPN-812; Test type: Superiority; p = 0.0063, Regression, Logistic; Risk Difference (RD) = 14.5, 95% CI 2-sided [4.3 to 24.6]
Statistical Analysis 2: Comparison: Placebo vs 200mg SPN-812; Test type: Superiority; p < 0.0001, Regression, Logistic; Risk Difference (RD) = 21.5, 95% CI 2-sided [11.3 to 31.6]

6. Secondary Outcome: Effect of SPN-812 Assessed by Parenting Stress Index, Fourth Edition, Short Form (PSI-4-SF)
Description: An additional secondary endpoint was the change from baseline in Parenting Stress Index, Fourth Edition, Short Form (PSI-4-SF) Total score at Week 6 (End of Study). The PSI-4 questionnaire evaluates the magnitude of stress in the parent-child relationship based on the parent's perception of the child's characteristics, the personal characteristics of the parent, and the interaction between the parent and the child. The PSI-4-SF was developed for parents of children ages 1 month to 12 years. The PSI-4-SF consists of 36 items divided into three domains: parental distress, parent-child dysfunctional interaction, and difficult child. Each item is rated on a 5-point Likert scale, where SD=Strongly Disagree, D=Disagree, NS=Not Sure, A=Agree, and SA=Strongly Agree. The total score ranges between 90 and 450; higher total scores indicate higher levels of stress. Lower change from baseline total scores (<0) represent better outcome.
Time Frame: Baseline and Week 6 (End of Study)
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | 100mg SPN-812 | 200mg SPN-812
Number analyzed (Participants) | 155 | 147 | 158
score on a scale | -8.5 (1.61) | -8.5 (1.63) | -10.1 (1.58)
Statistical Analysis 1: Comparison: Placebo vs 100mg SPN-812; Test type: Superiority; p = 0.9974, ANCOVA; Least Square Mean Difference = 0.00, 95% CI 2-sided [-4.5 to 4.5], Standard Error of Mean 1.63
Statistical Analysis 2: Comparison: Placebo vs 200mg SPN-812; Test type: Superiority; p = 0.4557, ANCOVA; Least Square Mean Difference = -1.7, 95% CI 2-sided [-6.1 to 2.7], Standard Error of Mean 2.26

7. Secondary Outcome: Effect of SPN-812 Assessed by the Hyperactivity/Impulsivity Subscale and the Inattention Subscale of the Attention-Deficit/Hyperactivity Disorder Rating Scale, 5th Edition (ADHD-RS-5)
Description: An additional secondary endpoint was the change from baseline in the Attention-Deficit/Hyperactivity Disorder Rating Scale, 5th Edition (ADHD-RS-5) Hyperactivity/Impulsivity subscale score and Inattention subscale score at Week 6 (End of Study). The ADHD-RS-5 is an ADHD-specific rating scale designed and validated to assess current ADHD symptomatology. The scale consists of 18 items that directly correspond to the 18 DSM-5 symptoms of ADHD, including 9 items for the Hyperactivity/Impulsivity subscale and 9 items for the Inattention subscale. Each item is rated on a 4-point Likert-type scale from 0 (never or rarely) to 3 (very often). Each subscale score is calculated by adding the responses of all respective 9 items (range: 0-27; the higher the subscale score, the more severe the Hyperactivity/Impulsivity or Inattention symptoms). Lower change from baseline subscale scores (<0) represent a better outcome.
Time Frame: Baseline and Week 6 (End of Study)
Population: as for baseline characteristics
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | 100mg SPN-812 | 200mg SPN-812
Number analyzed (Participants) | 155 | 147 | 158
score on a scale
  Inattention subscale | -5.7 (0.60) | -8.6 (0.62) | -9.2 (0.60)
  Hyperactivity/impulsivity Subscale | -5.5 (0.59) | -8.0 (0.60) | -8.7 (0.58)
Statistical Analysis 1: Comparison: Placebo vs 100mg SPN-812; This statistical analysis pertains to the Inattention subscale score; Test type: Superiority; p = 0.0006, ANCOVA; Least Square Mean Difference = -2.9, 95% CI 2-sided [-4.6 to -1.2], Standard Error of Mean 0.85
Statistical Analysis 2: Comparison: Placebo vs 200mg SPN-812; This statistical analysis pertains to the Inattention subscale score; Test type: Superiority; p < 0.0001, ANCOVA; Least Square Mean Difference = -3.5, 95% CI 2-sided [-5.2 to -1.9], Standard Error of Mean 0.83
Statistical Analysis 3: Comparison: Placebo vs 100mg SPN-812; This analysis pertains to the Hyperactivity/Impulsivity subscale score; Test type: Superiority; p = 0.0026, ANCOVA; Least Square Mean Difference = -2.5, 95% CI 2-sided [-4.1 to -0.9], Standard Error of Mean 0.83
Statistical Analysis 4: Comparison: Placebo vs 200mg SPN-812; This analysis pertains to the Hyperactivity/Impulsivity subscale score; Test type: Superiority; p < 0.0001, ANCOVA; Least Square Mean Difference = -3.2, 95% CI 2-sided [-4.8 to -1.7], Standard Error of Mean 0.81

8. Secondary Outcome: Effect of SPN-812 Assessed by Conners 3 - Self Report Short Form (C3-SRS)
Description: An additional secondary endpoint was the change from baseline in the Conners 3rd Edition - Self Report Short Form (C3-SRS) Composite T score at Week 6 (End of Study). The Conners 3rd Edition is a focused diagnostic tool for assessment of ADHD and associated learning, behavior, and emotional problems in children 6 to 18 years of age. The C3-SRS, which is only validated in children/adolescents 8-18 years of age, is comprised of 41 items with subsets of items related to five content scales: inattention, hyperactivity/impulsivity, learning problems, aggression and family relations. The subject rates himself/herself on the first 39 items of C3-SRS using a 4-point Likert scale (0-3; where 0=not at all true [never, seldom] and 3=very much true [very often, very frequently] based on past month; the last 2 items are fill-in-the-blank and do not contribute to the raw score(s). Raw scores are converted to T-scores. Lower change from baseline T-scores (<0) represent a better outcome.
Time Frame: Baseline and Week 6 (End of Study)
Population: Intent-to-Treat (ITT) Population: The ITT population includes subjects who were randomized, took at least one dose of study medication, have a baseline Attention-Deficit/Hyperactivity Disorder Rating Scale, 5th Edition (ADHD-RS-5) assessment and have at least one post-baseline ADHD-RS-5 assessment. There is a lower 'N' for this scale because the scale was only completed by subjects 8 to 11 years of age, since this specific scale is only validated in children 8-18 years of age.
Measure: Least Squares Mean (Standard Error); unit: T-score
Arm/Group | Placebo | 100mg SPN-812 | 200mg SPN-812
Number analyzed (Participants) | 100 | 102 | 107
T-score | -3.5 (0.85) | -5.3 (0.84) | -4.6 (0.83)
Statistical Analysis 1: Comparison: Placebo vs 100mg SPN-812; Test type: Superiority; p = 0.1292, ANCOVA; Least Square Mean Difference = -1.8, 95% CI 2-sided [-4.2 to 0.5], Standard Error of Mean 1.20
Statistical Analysis 2: Comparison: Placebo vs 200mg SPN-812; Test type: Superiority; p = 0.3447, ANCOVA; Least Square Mean Difference = -1.1, 95% CI 2-sided [-3.4 to 1.2], Standard Error of Mean 1.19

9. Secondary Outcome: Effect of SPN-812 Assessed by Categorical Clinical Global Impression - Improvement (CGI-I) [the Percentage of Subjects Who Were 'Improved"]
Description: An additional secondary endpoint was the percentage of subjects who were "improved" by visit; "improved" was defined as a subject who had a Clinical Global Impression - Improvement (CGI-I) score of 1 = "Very Much Improved" or 2 = "Much Improved". Values range from 0 to 100%. A higher percentage represents a greater number of subjects who were "improved".
Time Frame: Week 1, Week 2, Week 3, Week 4, Week 5, Week 6
Population: as for baseline characteristics
Measure: Number; unit: percentage of subjects
Arm/Group | Placebo | 100mg SPN-812 | 200mg SPN-812
Number analyzed (Participants) | 155 | 147 | 158
percentage of subjects
  Week 1 | 9.1 | 23.9 | 10.9
  Week 2 | 18.9 | 30.5 | 31.8
  Week 3 | 26.7 | 40.7 | 38.9
  Week 4 | 29.3 | 46.5 | 48.2
  Week 5 | 30.7 | 46.3 | 48.1
  Week 6 | 29.5 | 45.0 | 50.7
Statistical Analysis 1: Comparison: Placebo vs 100mg SPN-812; This analysis pertains to Week 1 of treatment; Test type: Superiority; p = 0.0005, Chi-squared
Statistical Analysis 2: Comparison: Placebo vs 100mg SPN-812; This analysis pertains to Week 2 of treatment; Test type: Superiority; p = 0.0212, Chi-squared
Statistical Analysis 3: Comparison: Placebo vs 100mg SPN-812; This analysis pertains to Week 3 of treatment; Test type: Superiority; p = 0.0115, Chi-squared
Statistical Analysis 4: Comparison: Placebo vs 100mg SPN-812; This analysis pertains to Week 4 of treatment; Test type: Superiority; p = 0.0027, Chi-squared
Statistical Analysis 5: Comparison: Placebo vs 100mg SPN-812; This analysis pertains to Week 5 of treatment; Test type: Superiority; p = 0.0066, Chi-squared
Statistical Analysis 6: Comparison: Placebo vs 100mg SPN-812; This analysis pertains to Week 6 of treatment; Test type: Superiority; p = 0.0065, Chi-squared
Statistical Analysis 7: Comparison: Placebo vs 200mg SPN-812; This analysis pertains to Week 1 of treatment; Test type: Superiority; p = 0.5826, Chi-squared
Statistical Analysis 8: Comparison: Placebo vs 200mg SPN-812; This analysis pertains to Week 2 of treatment; Test type: Superiority; p = 0.0099, Chi-squared
Statistical Analysis 9: Comparison: Placebo vs 200mg SPN-812; This analysis pertains to Week 3 of treatment; Test type: Superiority; p = 0.0225, Chi-squared
Statistical Analysis 10: Comparison: Placebo vs 200mg SPN-812; This analysis pertains to Week 4 of treatment; Test type: Superiority; p = 0.0008, Chi-squared
Statistical Analysis 11: Comparison: Placebo vs 200mg SPN-812; This analysis pertains to Week 5 of treatment; Test type: Superiority; p = 0.0020, Chi-squared
Statistical Analysis 12: Comparison: Placebo vs 200mg SPN-812; This analysis pertains to Week 6 of treatment; Test type: Superiority; p = 0.0002, Chi-squared

ADVERSE EVENTS:
Time Frame: 6 weeks
Description: Number of subjects is based on the Safety Population (defined as subjects who were randomized and took at least one dose of study medication)
Groups:
- Placebo: Placebo oral capsule
  Treatment A: Placebo administered once daily
- 100mg SPN-812: SPN-812 oral capsule
  Treatment B: 100mg SPN-812 administered once daily and compared to placebo
- 200mg SPN-812: SPN-812 oral capsule
  Treatment C: 200mg SPN-812 administered once daily and compared to placebo
Arm/Group | Placebo | 100mg SPN-812 | 200mg SPN-812
All-Cause Mortality (participants affected / at risk) | 0/159 | 0/154 | 0/161
Serious Adverse Events (participants affected / at risk) | 0/159 | 2/154 | 1/161
Other Adverse Events (participants affected / at risk) | 15/159 | 54/154 | 70/161
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=159) | 100mg SPN-812 (N=154) | 200mg SPN-812 (N=161)
Pyromania (Psychiatric disorders) | 0 | 1 | 0
Conduct disorder (Psychiatric disorders) | 0 | 1 | 0
Appendicitis (Gastrointestinal disorders) | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=159) | 100mg SPN-812 (N=154) | 200mg SPN-812 (N=161)
Headache (Nervous system disorders) | 6 | 15 | 16
Somnolence (Nervous system disorders) | 3 | 16 | 15
Decreased appetite (Metabolism and nutrition disorders) | 0 | 8 | 14
Vomiting (Gastrointestinal disorders) | 3 | 7 | 8
Nasopharyngitis (Infections and infestations) | 3 | 5 | 8
Sedation (Nervous system disorders) | 0 | 3 | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2018-08-22): https://cdn.clinicaltrials.gov/large-docs/30/NCT03247530/Prot_000.pdf
  • Statistical Analysis Plan (2018-10-17): https://cdn.clinicaltrials.gov/large-docs/30/NCT03247530/SAP_001.pdf